CLINICAL TRIAL: NCT06076291
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of SG1827 in Subjects With Advanced Solid Tumors
Brief Title: An Open-label Study of SG1827 in Subjects With Advanced Solid Tumors
Acronym: CSG-1827-101
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Sumgen Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSG-1827-101
Record Dates: First submitted 2023-09-24; First posted 2023-10-10 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SG1827 (Experimental): SG1827 monotherapy intravenous (IV) infusion - administered every three weeks (Q3W)
  Interventions: Drug: SG1827

INTERVENTIONS:
Drug: SG1827 — PhaseⅠa will use an accelerated titration and Bayesian optimal interval (AT-BOIN) design with 7 dose cohorts: 0.02mg/kg, 0.2mg/kg, 1mg/kg, 3mg/kg, 6mg/kg, 10mg/kg, and 15mg/kg by IV infusion. Accelerated titration (1 patient) will be only applied to the first cohort.

SUMMARY:
This is a Phase I, open-label, dose escalation and dose expansion study to Evaluate the Safety, Tolerability and Preliminary Efficacy of SG1827 in subjects with Advanced Solid Tumors, refractory or resistant to standard therapy, or without available standard or curative therapy.

DETAILED DESCRIPTION:
After a screening period of up to 28 days for each study phase, qualified patients will be enrolled to receive their assigned dose of SG1827, administered every three weeks (Q3W), until disease progression, intolerable toxicity or others, whichever occurs first.

The study consists of a dose escalation phase (Phase 1a) to determine the maximum tolerated dose (MTD), or recommended Phase 2 dose (RP2D) for SG1827 as a single agent, and a dose expansion phase (Phase 1b) in subjects with specific tumor types which will characterize treatment of SG1827 as a single agent at the MTD or RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign the informed consent form (ICF).
2. Age ≥18 years.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
4. Life expectancy ≥3 months.
5. Histologically or cytologically documented advanced or metastatic solid tumors that is refractory/relapsed to standard therapies, or for which no effective standard therapy is available. In the dose-expansion cohorts (Phase 1b), histologically or cytologically confirmed selected advanced solid tumors.
6. Subject must have at least one measurable lesion according to RECIST Version1.1.
7. Adequate organ function.
8. Toxicity caused by prior anti-tumor therapy recovered to Grade 0 to 1 (CTCAE 5.0).
9. Female patients of childbearing potential and male patients whose female partners are of childbearing potential need to use at least one approved contraceptive (e.g., intrauterine device, pill, or condom) during study treatment and for at least 5 months (150 days) after the last dose; female patients of childbearing potential must have a negative blood human chorionic gonadotropin (HCG) test within 7 days prior to dosing and must not be lactating.
10. Male patients must refrain from donating sperm from the time the ICF is signed until at least 5 months after the last dose.

Exclusion Criteria:

1. Subjects with symptomatic central nervous system metastatic lesions; presence of metastases to the brainstem or meninges, spinal cord metastases or compression. Except the subjects who have been treated, be asymptomatic.
2. Active autoimmune disease requiring systemic therapy within the past 2 years (e.g., use of immunomodulatory drugs, corticosteroids, or immunosuppressive medications); related replacement therapy is allowed (e.g., thyroid hormone, insulin, or physiologic corticosteroid replacement for renal or pituitary insufficiency).
3. Have received any of the following treatments or procedures:

   1. Prior treatment with any antitumor therapy targeting CTLA-4.
   2. Subjects received open surgery within 28 days prior to the first dose (except for surgeries for the purpose of biopsy).
   3. Subjects received systemic anticancer therapy (including chemotherapy, targeted therapy, hormonal therapy, immunotherapy and other experimental drugs) within 28 days or 5 drug half-lives (which occurs first) prior to the first dose, and all AEs have not returned to grade ≤1 (CTCAE 5.0).
   4. Subjects received curative radiotherapy within 28 days prior to the first dose; palliative radiotherapy is allowed if which occurs within 14 days prior to the first dose, and all AEs have not returned to grade ≤1 (CTCAE 5.0).
   5. Any live vaccine within 28 days prior to the first dose.
   6. Prior allogeneic organ grafting or allogeneic stem cell transplantation.
4. Subjects received systemic corticosteroids (equivalent dose > 10 mg/day of prednisone) or other immunosuppressive drugs within 14 days prior to the first dose or will receive during the study. Except topical or prophylactic treatment for non-autoimmune diseases.
5. Presence of active infection requiring antibiotic therapy within 30 days prior to the first dose, except for prophylaxis use.
6. Presence of cardiovascular system disease within 6 months prior to screening that meets any of the following:

   1. Cardiac function: congestive heart failure of New York Heart Association (NYHA) class III or IV; left ventricular ejection fraction <50%.
   2. Clinically significant cardiac disease or surgery , including myocardial infarction, unstable angina pectoris, coronary/peripheral artery bypass, etc.
   3. QTcF >450 ms (corrected QT interval with Fridericia formula); history of clinically significant ventricular arrhythmias (e.g., sustained ventricular tachycardia, ventricular fibrillation, tip-twist ventricular tachycardia); history or family history of congenital long QT syndrome; arrhythmias requiring antiarrhythmic drug therapy (patients with atrial fibrillation with controllable heart rate 1 month prior to the first dose of the investigational drug may be enrolled).
   4. History of arterial thrombosis, deep venous thrombosis and pulmonary embolism.
7. Hyperglycaemia or Hypertension that has not been effectively controlled after standard treatment.
8. Patients with active hepatitis B or C, or HIV antibody positive.
9. Known history of Grade 3 to 4 hypersensitivity reactions to any biological product, history of life threatening hypersensitivity reactions, or known hypersensitivity to components of SG1906 drug product.
10. History of interstitial lung disease or non-infectious pneumonitis except for those induced by radiation therapies.
11. Presence of body fluid (hydrothorax, ascites, pericardial effusion, etc.) requiring local treatment or repeated drainage.
12. Immune-related adverse effects leading to permanent discontinuation during previous antineoplastic immunotherapy.
13. Subjects with unhealed wounds.
14. Subjects with high risk of bleeding.
15. Subjects with other malignant solid tumors (except for cured defined tumors) within 5 years prior to the first dose.
16. Any other condition that, in the opinion of the Investigator, may lead to inappropriate participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Through study completion, an average of one year
  Number and percentage of AEs which is calculated by worst CTCAE grade by CTCAE 5.0
MTD/MAD/ RP2D | Through study completion, an average of one year
  MTD/MAD/RP2D will be determined based on the DLTs and safety data.

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Cmax | Through study completion, an average of one year
  Cmax to maximum drug concentrationadministration
Pharmacokinetics (PK):limination half-life (T1/2) | Through study completion, an average of one year
  limination half-life (T1/2) of the drug after administration.
PD endpoints: cytokine levels | Through study completion, an average of one year
  including but not limited to tumor necrosis factor (TNF)-α, interferon gamma (IFN-γ), interleukin (IL)-2, IL-4, IL-6, IL-8, IL-10, IL-1β.
Immunogenicity endpoints: | Through study completion, an average of one year
  levels of anti-drug antibodies (ADAs) and neutralizing antibodies (tested in ADA-positive samples only).
Efficacy endpoints: | Through study completion, an average of one year
  objective response rate (ORR),

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The Affiliated Hospital of USTC, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhenzhou, Henan
  - The Affiliated Cancer Hospital of Xiangya School of Medicine, Central South University, Changsha, Hunan
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No